CLINICAL TRIAL: NCT05242926
Title: Absorption and Excretion of Docetaxel (as ModraDoc 006 Tablets) After Oral Administration in Combination With Ritonavir
Brief Title: Absorption and Excretion of Oral Docetaxel
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Pending further development
Sponsor: Modra Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N16AED
Record Dates: First submitted 2017-07-17; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Intervention Model Description: Six evaluable patients will receive bidaily dosing on day 1 of week 1, whereafter collection of plasma, faeces and urine samples will take place until 168 hours after the first dosing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ModraDoc006/r (Experimental): Six evaluable patients will be included for collection of plasma, faeces and urine samples during 168 hours after one day of bi-daily dosing (30/20 mg) of ModraDoc006 in combination with ritonavir.
  Interventions: Drug: ModraDoc006/r

INTERVENTIONS:
Drug: ModraDoc006/r — One time bi-daily dosing (30/20 mg) of ModraDoc006 in combination with ritonavir 100 mg tablets
  Other Names: oral docetaxel formulation

SUMMARY:
This is an open-label, phase I study to investigate the influence of the bi-daily weekly dosing of ModraDoc006/ritonavir on the absorption and excretion of docetaxel in patients with advanced solid tumours.

The pharmacokinetics, absorption and excretion of docetaxel will be investigated during the study.

Patients will receive 30 mg in the morning / 20 mg in the afternoon ModraDoc006 with BID 100 mg ritonavir in a fasted condition (i.e. at least 1 hour before or 2 hours after any food assumption), followed by collection of plasma, faeces and urine samples.

DETAILED DESCRIPTION:
Oral administration of (anticancer) drugs has many advantages over the intravenous route. However, oral bioavailability of the docetaxel IV-formulation is low and variable. The bioavailability of docetaxel is limited due to metabolizing cytochrome P450 (CYP) enzymes, especially CYP3A, which are abundantly present in the gastrointestinal tract. Inhibition of CYP3A4 enzymes with ritonavir has proven to enhance the bioavailability of oral docetaxel in several pre-clinical and early clinical studies.

The Pharmacy of The Netherlands Cancer Institute has developed a new oral formulation of docetaxel (ModraDoc006), which contains a spray dried docetaxel powder resulting in an increased apparent solubility and therefore improved uptake from the gastrointestinal tract. The oral docetaxel ModraDoc006 tablet formulation, has been investigated in two phase I trials in combination with ritonavir. The combination of ModraDoc006/ritonavir resulted in a significantly increased bioavailability, reaching an exposure in terms of the area under plasma concentration-time curve (AUC) comparable to exposure observed after intravenous administration of weekly docetaxel at 35 mg/m2. Commonly observed toxicities in the phase I trials were nausea, diarrhea, fatigue, vomiting and alopecia, most being of grade 1-2.

The metabolism of docetaxel (as ModraDoc006) after oral administration in combination with ritonavir has not been investigated yet, nor have the routes of elimination been explored. Phase I clinical trials have focused on safety and pharmacokinetics of oral docetaxel after weekly once daily and bi-daily administration.

An absorption and excretion study after oral administration of a bi-daily dose of ModraDoc006/ritonavir can provide essential knowledge on the absorption, metabolism and excretion of this formulation of docetaxel. This knowledge can be used for further development. Using validated LC-MS/MS assays, docetaxel can be quantified in plasma, urine and faeces. Further analysis using a combination of chromatography, UV spectrometry and mass spectrometry may result in detection and quantification of its known metabolites M1, M2, M3 and M4 and as yet unidentified metabolites.

ELIGIBILITY:
Inclusion criteria

1. Histological or cytological proof of cancer.
2. Patients who might benefit from treatment with docetaxel, e.g. advanced breast, gastric, esophagus, bladder, ovarian cancer and non-small cell lung cancer, head and neck cancer, prostate cancer and carcinoma of unknown primary site.
3. Age ≥ 18 years.
4. Able and willing to give written informed consent.
5. WHO performance status of 0, 1 or 2.
6. Able and willing to undergo blood sampling, urine and faeces sampling for PK.
7. Able and willing to comply with the study protocol for the duration of the study.
8. Life expectancy ≥ 3 months.
9. Evaluable disease
10. Minimal acceptable safety laboratory values:

    1. ANC of ≥ 1.5 x 109/L
    2. Platelet count of ≥ 100 x 109/L
    3. Hepatic function as defined by serum bilirubine ≤ 1.5 x ULN, ASAT and ALAT ≤ 2.5 x ULN (or ≤ 5 ULN in case of liver metastases)
    4. Renal function as defined by serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min (by Cockcroft-Gault formula)
11. Negative pregnancy test (urine/serum) for female patients with childbearing potential.
12. No radio- or chemotherapy within 4 weeks prior to the first dose of ModraDoc006/r (palliative radiation on a limited field for pain control is allowed)
13. Able and willing to swallow oral medication.

Exclusion criteria

1. Patients with known alcoholism, drug addiction and/or psychotic disorders in the history that are not suitable for adequate follow up.
2. Women who are pregnant or breast-feeding.
3. Unreliable contraceptive methods. Both men and women enrolled in this trial must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are described in section 8.8.3 and include condom, sterilization and other barrier contraceptive measures preferably in combination with condoms).
4. Concomitant use of MDR and CYP3A modulating drugs, including but not limited to Ca2+-entry blockers (verapamil, dihydropyridines), cyclosporine, quinidine, quinine, tamoxifen, megestrol and grapefruit juice, concomitant use of HIV medications; other protease inhibitors, (non) nucleoside analogs, St. John's wort or macrolide antibiotics as erythromycin and clarithromycin. A washout period is established for all relevant drugs (see appendix VII).
5. Uncontrolled infectious disease or known HIV-1 or HIV-2 type infection.
6. Unresolved (>grade 1) toxicities of previous chemotherapy, excluding alopecia.
7. Bowel obstructions, motility disorders or previously performed extended abdominal surgery that may influence the absorption of drugs.
8. Neurologic disease that may render a patient at increased risk for peripheral or central neurotoxicity.
9. Pre-existing neuropathy greater than CTC grade 1.
10. Patients with symptomatic brain metastases or with leptomeningeal metastases. Patients with brain metastases are allowed if they received adequate treatment, are asymptomatic in the absence of corticosteroid therapy and anticonvulsant therapy for at least 6 weeks. Radiotherapy for brain metastasis must have been completed at least 6 weeks prior to start of study treatment. Brain metastasis must be stable with verification by imaging (e.g. brain MRI or CT completed at screening).
11. Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The absorption of oral docetaxel | Pharmacokinetic sampling during 48 hours - 168 hours
  Using validated LC-MS/MS assays, docetaxel can be quantified in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Serena Marchetti, MD/PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No